CLINICAL TRIAL: NCT06453304
Title: Clinical Investigation of the Effectiveness of Glycyrrhizin as Intracanal Medication in Root Canal Disinfection and Inflammatory Cytokines
Brief Title: Effectiveness of Glycyrrhizin as Intracanal Medication in Root Canal Disinfection and Inflammatory Cytokines
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Intracanal medication
Record Dates: First submitted 2024-05-27; First posted 2024-06-11 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Intracanal Medication
Keywords: Glycirrhizin cytokines antibacterial
MeSH Terms: interventions — Calcium Hydroxide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Calcium Hydroxide (Active Comparator)
  Interventions: Drug: Calcium Hydroxide
- Leddermix (Active Comparator)
  Interventions: Drug: Leddermix
- Glycirrhizin (Active Comparator)
  Interventions: Drug: Glycirrhizin

INTERVENTIONS:
Drug: Calcium Hydroxide — Intracanal medication
  Arms: Calcium Hydroxide
Drug: Leddermix — Intracanal medication
  Arms: Leddermix
Drug: Glycirrhizin — Intracanal medication
  Arms: Glycirrhizin

SUMMARY:
The objective of this study is to investigate "clinically" the effectiveness of Glycyrrhizin based intracanal medication compared to the commonly used intracanal medicaments (calcium hydroxide Ca(OH)2 and Ledermix) on the levels of bacteria and inflammatory cytokines in root canals and periradicular tissues of teeth with apical periodontitis.

DETAILED DESCRIPTION:
Periodontitis is a dynamic inflammatory process located at the periapical region, the type of immune-inflammatory response to periapical periodontitis is determined by a network of chemical mediators produced by immune cells in response to the stimulus caused by the action of microorganisms and/or virulence factors. This may result in damage to the tissues and in the development of endodontic signs and symptoms (1-3).

In infected root canals, the destruction of periapical tissues is mediated by tumor necrotizing factor (TNF-α) and interleukin-1β (IL-1β) that appears to be directly related to high levels of infectious content present in the root canal (4). Arachidonic acid metabolism plays a key role in many inflammatory diseases, one of its products is the prostaglandin E2 (PGE2) which has been also shown to potentially stimulate bone resorption and to inhibit reparative bone formation in vitro and in vivo (5). Particularly, IL-1β, TNF-α, and PGE2 have been detected in periapical tissues (6-9), being considered as an important inflammatory biomarker in the periapical disease (1, 2, 5, 7, 10).

To identify a specific inflammatory mediator as a diagnostic marker of disease status, the mediator should not only be present or elevated in disease and absent or low in health, but it should also longitudinally increase during active disease progression and subside following therapy (5).

Although instrumentation may be assumed to be of greater importance in the clinical practice, the use of intracanal medication has been proven to optimize the root canal disinfection (11-14). As root canal medicaments can come in direct contact with periapical tissues, in addition to having good antibacterial ability and being biocompatible, so a wide variety of intracanal medications have been proposed. In selecting root canal medicaments, it is necessary to consider their therapeutic benefits against their potential cytotoxic effects. Ideal root canal medicaments should have strong antibacterial properties and minimal cytotoxic effect on the host tissues (11-16).

Calcium hydroxide (Ca(OH)2) has been used extensively in dentistry since the 1920s (17). Today, it is still the most commonly used endodontic medicament throughout the world(18).Ca(OH)2 also inactivates lipopolysaccharide so it can assist in periapical tissue repair (19).

Corticosteroids have also shown to interfere with the repair process. This interference includes an inhibition of fibroblastic proliferation and a decrease in polymorphonuclear leukocyte locomotion. In addition, corticosteroids interfere with the immune response, which could disseminate bacteria leading to infectious disease. Considering these potential pitfalls, some investigators have advocated supplemental use of an antibiotic to help control infection. As a result, ledermix paste was used where it consists of both a corticosteroid "triamcinolone" and an antibiotic "dimethyl chlortetracycline" (20, 21).

Herbs have been used in clinical medicine for thousands of years. Recently researchers have been able to employ scientific methods to prove the efficacy of many of these herbs and to provide a better understanding of their mechanisms of action (22).

Glycyrrhiza glabra which is known as licorice belonging to the Fabaceae, is native to southern Europe and parts of Asia including Iran (23). Licorice roots have been used as a remedy for cough, constipation, menopausal hot flashes, peptic ulcer, and viral diseases (24). Licorice contains more than 20 triterpenoids and nearly 300 flavonoids. Among them, glycyrrhizin, 18 β-glycyrrhetinic acid, liquiritigenin, licochalcone A, licochalcone E and glabridin are the main active components which possess antimicrobial, antioxidant and anti-inflammatory activities (25-27). Badr et al. (28) reported that Licorice extract either separately or as Liquorice/Ca(OH)2 mixture had a potent bactericidal effect against Enterococcus faecalis and retained compatibility with fibroblasts in tissue culture compared to the commonly used root canal medicament Ca(OH)2.

Glycyrrhizin (an oleanane-type triterpenoid glucuronide), the main active and important constituent in licorice, is 50 times sweeter than sugar (29) and is used in large quantities as a well-known natural sweetener and as a pharmaceutical (30). It is a conjugate of two molecules of glucuronic acid and glycyrrhetinic acid and is found chiefly in roots and stolons but not in aerial parts (31). Glycyrrhizin possesses anti-allergic (32), anti- diabetic (33), anti-inflammatory (34), anti-ocular hypertension (35), immune-modulatory (36), anti-cholestasis (37), hepatoprotective (38) and neuroprotective pharmacological activities (39). It also has protective effect on the respiratory system (40).

So based on the above mentioned data, it is believed to be of interest to investigate clinically the use of Glycyrrhizin as an intracanal medication.

ELIGIBILITY:
Inclusion Criteria:

* Single-rooted with pulp necrosis and apical periodontitis.

Exclusion Criteria:

* Receiving antibiotic treatment within the preceding 3 months.
* Reporting systemic disease.
* Teeth that could not be isolated with rubber dam.
* Teeth with periodontal pockets deeper than 3 mm.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2022-03-20 (Actual); Primary Completion 2024-06-05 (Actual); Study Completion 2024-07-10 (Estimated)

PRIMARY OUTCOMES:
counting the number of colonies forming units of bacterial cells | up to 7 months
  Microbiology cell culturing (manual counting technique to the bacterial cells)

OTHER OUTCOMES:
using enzyme-linked immunosorbent assay (ELISA test) to measure the amount of Inflammatory Cytokines (TNF-α), (IL-1β) and (PG2) | 25 weeks
  ELISA test to measure the amount of tumor necrotizing factor (TNF-α), interleukin 1β(IL-1β) and prostaglandin E2 (PG2)

CONTACTS AND LOCATIONS:
Overall Officials: Amany Badr, Prof, Study Chair — Faculty of Dentistry Mansoura University; Youssry Elhawary, Prof, Study Director — Faculty of Dentistry Mansoura University; Ghada Abdelrazik, Dr, Study Director — Faculty of Dentistry Mansoura University
Locations (1):
- Alaa Reda Mohamed Eltantawi, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Martinho FC, Chiesa WM, Leite FR, Cirelli JA, Gomes BP. Antigenic activity of bacterial endodontic contents from primary root canal infection with periapical lesions against macrophage in the release of interleukin-1beta and tumor necrosis factor alpha. J Endod. 2010 Sep;36(9):1467-74. doi: 10.1016/j.joen.2010.06.012. PMID 20728711
- [Background] Vianna ME, Horz HP, Conrads G, Zaia AA, Souza-Filho FJ, Gomes BP. Effect of root canal procedures on endotoxins and endodontic pathogens. Oral Microbiol Immunol. 2007 Dec;22(6):411-8. doi: 10.1111/j.1399-302X.2007.00379.x. PMID 17949345
- [Background] Athanassiadis B, Abbott PV, Walsh LJ. The use of calcium hydroxide, antibiotics and biocides as antimicrobial medicaments in endodontics. Aust Dent J. 2007 Mar;52(1 Suppl):S64-82. doi: 10.1111/j.1834-7819.2007.tb00527.x. PMID 17546863
- [Background] Tang G, Samaranayake LP, Yip HK. Molecular evaluation of residual endodontic microorganisms after instrumentation, irrigation and medication with either calcium hydroxide or Septomixine. Oral Dis. 2004 Nov;10(6):389-97. doi: 10.1111/j.1601-0825.2004.01015.x. PMID 15533217
- [Background] Badr AE, Omar N, Badria FA. A laboratory evaluation of the antibacterial and cytotoxic effect of Liquorice when used as root canal medicament. Int Endod J. 2011 Jan;44(1):51-8. doi: 10.1111/j.1365-2591.2010.01794.x. Epub 2010 Aug 31. PMID 20812941
- [Background] van der Sluis LW, Versluis M, Wu MK, Wesselink PR. Passive ultrasonic irrigation of the root canal: a review of the literature. Int Endod J. 2007 Jun;40(6):415-26. doi: 10.1111/j.1365-2591.2007.01243.x. Epub 2007 Apr 17. PMID 17442017
- [Result] Martinho FC, Chiesa WM, Leite FR, Cirelli JA, Gomes BP. Antigenicity of primary endodontic infection against macrophages by the levels of PGE(2) production. J Endod. 2011 May;37(5):602-7. doi: 10.1016/j.joen.2010.12.005. Epub 2011 Mar 5. PMID 21496656